CLINICAL TRIAL: NCT01982253
Title: A Phase 2 Randomized, Placebo-Controlled, Double-Blind Parallel-Group, Multicenter Study to Evaluate the Glycemic Effects and Safety of Fasiglifam 25 mg Twice Daily and 50 mg Once Daily on Glycemic Control in Subjects With Type 2 Diabetes
Brief Title: Fasiglifam 25 mg BID vs 50 mg QD
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to potential concerns about liver safety (See Detailed Description)
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-875_203; 2013-000886-35 (EudraCT Number); U1111-1146-1263 (Registry Identifier: WHO Unique Trial Number)
Record Dates: First submitted 2013-11-05; First posted 2013-11-13 (Estimated); Results first posted 2016-10-07 (Estimated); Last update posted 2016-10-07 (Estimated); Status verified 2016-08

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Drug therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — TAK-875

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Fasiglifam placebo-matching tablets, orally, twice daily for up to 12 weeks.
  Interventions: Drug: Placebo to fasiglifam
- Fasiglifam 25 mg BID (Experimental): Fasiglifam 25 mg tablets, orally, twice daily (BID) for up to 12 weeks.
  Interventions: Drug: Fasiglifam
- Fasiglifam 50 mg QD +Placebo QD (Experimental): Fasiglifam 50 mg tablets, orally once daily (QD) and fasiglifam placebo-matching tablets, orally, once daily for up to 12 weeks.
  Interventions: Drug: Fasiglifam; Drug: Placebo to fasiglifam

INTERVENTIONS:
Drug: Fasiglifam — Fasiglifam tablets
  Other Names: TAK-875
  Arms: Fasiglifam 25 mg BID; Fasiglifam 50 mg QD +Placebo QD
Drug: Placebo to fasiglifam — Fasiglifam placebo-matching tablets
  Arms: Fasiglifam 50 mg QD +Placebo QD; Placebo

SUMMARY:
To evaluate the efficacy of fasiglifam 25 mg twice daily (BID) and fasiglifam 50 mg once daily (QD) on glycemic control in adults with type 2 diabetes who are inadequately controlled on diet and exercise alone.

DETAILED DESCRIPTION:
The drug being tested in this study is called fasiglifam. Fasiglifam is being tested to treat people who have diabetes. This study will look at glycemic control in people who take fasiglifam.

The study will enroll approximately 400 patients. Participants will be randomly assigned (by chance) to one of the three treatment groups-which will remain undisclosed to the patient and study doctor during the study (unless there is an urgent medical need):

* Fasiglifam 25 mg twice a day
* Fasiglifam 50 mg once daily
* Placebo (dummy inactive pill) - this is a tablet that looks like the study drug but has no active ingredient.

All participants will be asked to take one tablet twice each day throughout the study. All participants will be asked to record any time they have symptoms of hypoglycemia in a diary.

This multi-center trial will be conducted worldwide. The overall time to participate in this study is 18 weeks. Participants will make 9 visits to the clinic.

Due to potential concerns about liver safety, on balance, the benefits of treating patients with fasiglifam (TAK-875) do not outweigh the potential risks.

For this reason, Takeda has decided voluntarily to terminate the development activities for fasiglifam.

ELIGIBILITY:
Inclusion Criteria:

1. In the opinion of the investigator, the participant is capable of understanding and complying with protocol requirements.
2. The participant or, when applicable, the participant's legally acceptable representative signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures.
3. Is male or female and 18 years of age or older with a historical diagnosis of Type 2 Diabetes Mellitus (T2DM).
4. Has a glycosylated hemoglobin (HbA1c) level ≥7.0% and ≤10.0% and fasting plasma glucose (FPG) ≤270 mg/dL (15.0 mmol/L) at Screening Visit.
5. Has been treated with diet and exercise but has not received treatment with antidiabetic agents within 12 weeks prior to Screening Visit (Exception: if a patient has received other antidiabetic therapy for ≤7 days in total within the 2 months prior to Screening Visit).
6. Has a body mass index (BMI) ≤45 kg/m^2 at Screening.
7. If regularly using other, non-excluded medications, must be on a stable dose for at least 4 weeks prior to Screening Visit. However, as needed (PRN) use of prescription or over-the-counter medications is allowed at the discretion of the investigator.
8. Is able and willing to monitor glucose with a home glucose monitor and consistently record his or her own blood glucose concentrations and complete subject diaries.
9. A female of childbearing potential who is sexually active with a non-sterilized male partner agrees to routinely use adequate contraception from signing of the informed consent throughout the duration of the study and for 30 days after the last dose of study drug.

Exclusion Criteria:

1. Has received any investigational compound within 30 days prior to Screening Visit or has received an investigational anti-diabetic drug within the 3 months prior to Screening Visit.
2. Was randomized into a previous fasiglifam study.
3. Is an immediate family member, study site employee, or is in a dependent relationship with a study site employee who is involved in conduct of this study (eg, spouse, parent, child, sibling) or may consent under duress.
4. Has donated or received any blood products within 12 weeks prior to Screening or is planning to donate blood during the study.
5. Has a hemoglobin ≤12 g/dL (≤120 g/L) for males and ≤10 g/dL (≤100 g/L) for females at Screening.
6. Has a systolic blood pressure ≥160 mm Hg or diastolic pressure ≥95 mm Hg at Screening
7. Has a history of cancer that has been in remission for <5 years prior to Screening. A history of basal cell carcinoma or stage 1 squamous cell carcinoma of the skin is allowed.
8. Has alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) levels >2.0× upper limit of normal (ULN) at Screening.
9. Has a total bilirubin level greater than the ULN at Screening. Exception: if a patient has documented Gilbert's syndrome the patient will be allowed with an elevated bilirubin level per the investigator's discretion.
10. Has a serum creatinine ≥1.5 mg/dL (≥133μmol/L) (males) and ≥1.4 mg/dL (≥124 μmol/L) (females) and/or estimated glomerular filtration rate (eGFR) <60 mL/min/1.73m^2 at Screening.
11. Has uncontrolled thyroid disease as determined by the investigator.
12. Has a history of laser treatment for proliferative diabetic retinopathy within 6 months prior to Screening.
13. Had gastric banding, or gastric bypass surgery within one year prior to Screening.
14. Has a known history of infection with human immunodeficiency virus (HIV), hepatitis B virus, or hepatitis C virus.
15. Had coronary angioplasty, coronary stent placement, coronary bypass surgery, myocardial infarction, unstable angina pectoris, clinically significant abnormal electrocardiogram (ECG), cerebrovascular accident or transient ischemic attack within 3 months prior to or at Screening.
16. Has a history of hypersensitivity, allergies, or has had an anaphylactic reaction(s) to any component of fasiglifam.
17. Has a history of drug abuse (defined as illicit drug use) or a history of alcohol abuse within 2 years prior to Screening.
18. Received excluded medications prior to Screening Visit or is expected to receive excluded medication.
19. If female, is pregnant (confirmed by laboratory testing, ie, serum/urine human chorionic gonadotropin (hCG), in females of childbearing potential) or lactating or intending to become pregnant before, during, or within 1 month after participating in this study; or intending to donate ova during such time period.
20. The subject is unable to understand verbal or written English or any other language for which a certified translation of the approved informed consent is available.
21. The subject has any other physical or psychiatric disease or condition that in the judgment of the investigator may affect life expectancy or may make it difficult to successfully manage and follow the subject according to the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-10; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Senior Medical Director, Clinical Science, Study Director — Takeda
Locations (88):
- United States (47):
  - Goodyear, Arizona
  - Long Beach, California
  - Los Angeles, California
  - North Hollywood, California
  - Norwalk, California
  - Tustin, California
  - Boynton Beach, Florida
  - Coral Gables, Florida
  - Miami, Florida
  - Orlando, Florida
  - Pembroke Pines, Florida
  - Decatur, Georgia
  - Chicago, Illinois
  - Avon, Indiana
  - Franklin, Indiana
  - Greenfield, Indiana
  - Muncie, Indiana
  - Council Bluffs, Iowa
  - Topeka, Kansas
  - Lexington, Kentucky
  - Metairie, Louisiana
  - Flint, Michigan
  - Albuquerque, New Mexico
  - Charlotte, North Carolina
  - Greensboro, North Carolina
  - Mooresville, North Carolina
  - Morganton, North Carolina
  - Salisbury, North Carolina
  - Maumee, Ohio
  - Norman, Oklahoma
  - Corvallis, Oregon
  - Portland, Oregon
  - Harleysville, Pennsylvania
  - Levittown, Pennsylvania
  - Uniontown, Pennsylvania
  - Greer, South Carolina
  - Carrollton, Texas
  - Dallas, Texas
  - Edinburg, Texas
  - Houstan, Texas
  - Houston, Texas
  - New Braunfels, Texas
  - San Antonio, Texas
  - Spring, Texas
  - Salt Lake City, Utah
  - Burke, Virginia
  - Manassas, Virginia
- Bulgaria (7):
  - Byala
  - Pleven
  - Plovdiv
  - Rousse
  - Sevlievo
  - Sofia
  - Varna
- Poland (7):
  - Lodz
  - Oświęcim
  - Poznan
  - Rzeszów
  - Sobótka
  - Torun
  - Zgierz
- Romania (6):
  - Baia Mare
  - Bucharest
  - Cluj-Napoca
  - Iași
  - Oradea
  - Ploieşti
- Slovakia (12):
  - Bardejov
  - Bratislava
  - Dolný Kubín
  - Komárno
  - Levice
  - Lučenec
  - Nitra
  - Pezinok
  - Sabinov
  - Stropkov
  - Svidník
  - Štúrovo
- Taiwan (4):
  - Kaohsiung City
  - Taichung
  - Tainan
  - Taipei
- Ukraine (5):
  - Kharkiv
  - Kyiv
  - Simferopol
  - Ternopil
  - Vinnytsia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 5 investigative sites in the United States from 21 October 2013 to 31 January 2014.
Pre-assignment Details: Participants with a historical diagnosis of type 2 diabetes mellitus and inadequate glycemic control on diet and exercise alone were enrolled in 1 of 3 treatment groups, placebo, fasiglifam 25 milligram (mg) twice daily (BID) and fasiglifam 50 mg once daily (QD).
Groups:
- Placebo: Fasiglifam placebo-matching tablets, orally, twice daily for up to Day 47.
- Fasiglifam 25 mg BID: Fasiglifam 25 mg, tablets, orally, twice daily for up to Day 47.
- Fasiglifam 50 mg QD: Fasiglifam 50 mg, tablet, orally, once daily and fasiglifam- placebo matching tablet, orally, once daily for up to Day 47.
Period: Overall Study
Arm/Group | Placebo | Fasiglifam 25 mg BID | Fasiglifam 50 mg QD
Started | 2 | 4 | 4
Completed | 0 | 0 | 0
Not Completed | 2 | 4 | 4
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Study terminated by sponsor | 1 | 4 | 4

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who received at least 1 dose of double-blind study drug. Participants were analyzed according to the study drug they received.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Fasiglifam 25 mg BID | Fasiglifam 50 mg QD | Total
Number analyzed (Participants) | 2 | 4 | 4 | 10
Age, Customized [Number; unit: participants]
  18 to 64 years | 1 | 4 | 4 | 9
  65 to 84 years | 1 | 0 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 2 | 6
  Male | 1 | 1 | 2 | 4
Race/Ethnicity, Customized [Number; unit: participants]
  Black or African American | 1 | 0 | 1 | 2
  White | 1 | 4 | 3 | 8
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 1 | 3 | 1 | 5
  Not Hispanic or Latino | 1 | 1 | 3 | 5
Glycosylated Haemoglobin (HbA1c) [Number; unit: participants]
  Less than (<) 8.5 percent (%) | 2 [6.8 to 8.2] | 2 [6.8 to 9.3] | 3 [7.2 to 8.8] | 7
  Greater than or equal to (≥) 8.5 percent (%) | 0 | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in HbA1c at Week 12.
Description: The change in the value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at week 12 or final visit relative to baseline.
Time Frame: Baseline and Week 12
Population: In accordance with the SAP, due to the limited enrollment at the time of study termination, the summaries and statistical analyses of primary and secondary efficacy parameters originally intended and described in the protocol were not produced.
Arm/Group | Placebo | Fasiglifam 25 mg BID | Fasiglifam 50 mg QD
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Week 12
Description: The change between the FPG value collected at week 12 or final visit relative to baseline.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Arm/Group | Placebo | Fasiglifam 25 mg BID | Fasiglifam 50 mg QD
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started after the first dose of double-blind study drug and within 30 days after the last dose of double-blind study drug.
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Placebo | Fasiglifam 25 mg BID | Fasiglifam 50 mg QD
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 1/2 | 1/4 | 2/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=2) | Fasiglifam 25 mg BID (N=4) | Fasiglifam 50 mg QD (N=4)
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.